CLINICAL TRIAL: NCT02706795
Title: Dose-escalating Safety and Preliminary Efficacy of DaxibotulinumtoxinA for Injection in Cervical Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RT002-CL005
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Torticollis (Spasmodic)
Keywords: Cervical dystonia; Spasmodic torticollis
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

ARMS (1):
- daxibotulinumtoxinA (DAXI) for injection (Experimental): DAXI for injection
  Interventions: Biological: DaxibotulinumtoxinA

INTERVENTIONS:
Biological: DaxibotulinumtoxinA — Low, mid, and high dose sequential treatments of daxibotulinumtoxinA in dose-escalation safety and efficacy study

SUMMARY:
This is an open-label, dose-escalation study to assess the safety and preliminary efficacy of daxibotulinumtoxinA in subjects with isolated cervical dystonia (CD).

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for isolated cervical dystonia
* Has moderate severity with a baseline Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) - Total score of at least 20 and a TWSTRS-Severity subscale score or at least 15
* Has been using stable doses of focal dystonia medications for at least 3 months and willing to continue through end of study

Exclusion Criteria:

* Cervical dystonia attributable to an underlying etiology, such as traumatic torticollis or tardive torticollis; predominant retrocollis or anterocollis cervical dystonia
* Significant dystonia in other body areas, or is currently being treated with botulinum toxin for dystonia in other areas than isolated cervical dystonia
* Neurological abnormalities other than cervical dystonia
* History of severe dysphagia or aspiration, or current clinically significant swallowing disorder
* Previous neck surgery, phenol injection to the neck muscles, myotomy or denervation surgery in the neck/shoulder region, or intrathecal baclofen
* Marked limitation on passive range of motion that suggests contractures or other structural abnormality, e.g. cervical contractures or cervical spinal deformity
* Profound atrophy of cervical musculature
* Any neurological condition that may place the subject at increased risk with exposure to botulinum toxin type A, including peripheral motor neuropathic diseases such as amyotrophic lateral sclerosis and motor neuropathy, and neuromuscular junctional disorders such as Lambert-Eaton syndrome and myasthenia gravis
* Suboptimal efficacy response to any prior botulinum toxin type A product, when a previous treatment produced more optimal therapeutic response, as judged subjectively by the Investigator
* Previous treatment with any botulinum toxin product for any condition within the 6 months prior to Screening and during the study; presence of any blood coagulation disorder; or on anticoagulation treatment with international normalized ratio (INR) > 3.5

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12-07 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Improvement of dystonia as measured by change from baseline in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) - Total Score | Week 4

SECONDARY OUTCOMES:
Change from baseline in Toronto Western Spasmodic Torticollis Rating Scale(TWSTRS) - Total Score | Post-treatment: Weeks 2, 4, 6, 9, 12, 16, 20, 24
Change from baseline in TWSTRS subscale scores (Severity, Disability and Pain) | Post-treatment: Weeks 2, 4, 6, 9, 12, 16, 20, 24
Duration of effect based on number of weeks from treatment until return of symptoms that warrant treatment | Post-treatment: Weeks 2, 4, 6, 9, 12, 16, 20, 24
Percentage of treatment responders with at least a 20% reduction in the TWSTRS - Total score post-treatment | Weeks 2, 4, 6, 9, 12, 16, 20, 24
Patient-rated quality of life measurement based upon change from baseline of the Cervical Dystonia Impact Profile Scale (CDIP-58) | Post-treatment: Weeks 4, 6, 12, 16, 20, 24
Percentage of responders showing improvement on Clinical Global Impression of Change (CGIC) | Post-treatment: Weeks 2, 4, 6, 9, 12, 16, 20, 24

CONTACTS AND LOCATIONS:
Overall Officials: Nubia Kaba, Study Director — Sponsor GmbH
Locations (13):
- United States (13):
  - The Parkinson's & Movement Disorder Institute, Fountain Valley, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - University of Florida Center for Movement Disorders & Neurorestoration, Gainesville, Florida
  - Precision Research Organization, Miami Lakes, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kansas City Bone & Joint Clinic, Overland Park, Kansas
  - The NeuroMedical Center Clinic, Baton Rouge, Louisiana
  - Wake forest Baptist Health, Winston-Salem, North Carolina
  - Riverhills Healthcare, Inc., Cincinnati, Ohio
  - Coastal Neurology, Port Royal, South Carolina
  - Parkinson's Disease Center and Movement Disorder Clinic, Houston, Texas

REFERENCES:
- [Derived] Jankovic J, Truong D, Patel AT, Brashear A, Evatt M, Rubio RG, Oh CK, Snyder D, Shears G, Comella C. Injectable DaxibotulinumtoxinA in Cervical Dystonia: A Phase 2 Dose-Escalation Multicenter Study. Mov Disord Clin Pract. 2018 Apr 26;5(3):273-282. doi: 10.1002/mdc3.12613. eCollection 2018 May-Jun. PMID 30009213